CLINICAL TRIAL: NCT03588936
Title: Phase 1 Study of Nivolumab in Combination With Tocilizumab for Treatment of Patients With Relapsed Hematological Malignancies Post-allogeneic Transplant
Brief Title: Nivolumab and Tocilizumab for Relapsed Hematological Malignancy Post-allogeneic Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual and loss of funding.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nirav Shah, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO32525
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Acute Leukemia; Chronic Leukemia; Lymphoma; Myelodysplastic Syndromes
MeSH Terms: conditions — Lymphoma; Myelodysplastic Syndromes | interventions — Nivolumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab (0.25 mg/kg) and Tocilizumab (Experimental): Participant will receive tocilizumab 8 mg/kg IV (max dose 800 mg) on Day 0. On Day 1 participants will receive nivolumab IV (0.25 mg/kg based on dose escalation design).
  Nivolumab will be given every ~2 weeks for up to 4 doses and a second dose of Tocilizumab will be given on ~Day 29 on the same day as Dose # 3 of Nivolumab.
  Interventions: Drug: Nivolumab (.25 mg/kg); Drug: Tocilizumab
- Nivolumab (0.5 mg/kg) and Tocilizumab (Experimental): Participant will receive tocilizumab 8 mg/kg IV (max dose 800 mg) on Day 0. On Day 1 participants will receive nivolumab IV (0.5 mg/kg based on dose escalation design).
  Nivolumab will be given every ~2 weeks for up to 4 doses and a second dose of Tocilizumab will be given on ~Day 29 on the same day as Dose # 3 of Nivolumab.
  Interventions: Drug: Tocilizumab; Drug: Nivolumab (.5 mg/kg)

INTERVENTIONS:
Drug: Nivolumab (.25 mg/kg) — Participants will receive Nivolumab at one of two dose levels every 2 weeks for 4 treatments.
  Other Names: OPDIVO
  Arms: Nivolumab (0.25 mg/kg) and Tocilizumab
Drug: Tocilizumab — Participants will receive 2 doses of tocilizumab
  Other Names: ACTEMRA
Drug: Nivolumab (.5 mg/kg) — Participants will receive Nivolumab at one of two dose levels every 2 weeks for 4 treatments.
  Other Names: OPDIVO
  Arms: Nivolumab (0.5 mg/kg) and Tocilizumab

SUMMARY:
This is a phase 1, interventional single arm, open label, treatment study designed to evaluate the safety combination programmed cell death protein 1 (PD-1) and interleukin 6 (IL-6) inhibition in participants with relapsed disease post-allogeneic transplant.

DETAILED DESCRIPTION:
Study disease: Hematologic malignancies including, but not exclusive to,acute/chronic leukemia, lymphoma, and myelodysplastic syndrome that has relapsed after allogeneic transplant.

Study Rationale: Phase 1 Safety/Dose Finding Study: To determine the safety and maximum tolerated dose of Nivolumab in combination with Tocilizumab.

Study Agent Description:

Tocilizumab is a monoclonal antibody and immunosuppressant; specifically, tocilizumab is an IL-6 receptor antagonist.

Nivolumab is a human immunoglobulin G4 (IgG4) monoclonal antibody that binds to the PD-1 receptor of T cells blocking its interaction with PD-L1 and PD-L2, thereby enhancing T-cell proliferation and allowing the immune system to attack the tumor.

Number of Subjects: A maximum of 12 participants will be enrolled on this Phase 1 study.

Duration of Follow-up: Participants will be followed for up to one year post-treatment for survival and response.

Study Design: This is a 3 + 3 design. In a "3 + 3 design," three participants are initially enrolled into a given dose cohort. If there is no dose limiting toxicity (DLT) observed in any of these subjects, the trial proceeds to enroll additional subjects into the next higher dose cohort. If one subject develops a DLT at a specific dose, an additional three subjects are enrolled into that same dose cohort. Development of DLTs in more than one of six subjects in a specific dose cohort suggests that the maximum tolerated dose (MTD) has been exceeded, and further dose escalation is not pursued.

ELIGIBILITY:
Inclusion Criteria

1. Age≥18 years with hematological malignancies who have undergone allogeneic transplant for hematological malignancy and are ≥180 days post-transplant.
2. Relapsed disease post-allogeneic transplant defined as follows i. Acute or Chronic Leukemia or myelodysplastic or myeloproliferative disorders or natural killer (NK) cell neoplasms: Bone marrow (BM) with ≥5% disease involvement or peripheral blood evidence of overt relapse ii. Lymphoma: BM evidence of relapsed/persistent disease or PET/CT or CT evidence of persistent/progressive lymphadenopathy consistent with active lymphoma. Active disease defined as nodal lesions ≥ 20 mm in the long axis or extranodal lesions≥10 mm in long and short axis or bone marrow involvement that is biopsy proven
3. Karnofsky performance status ≥70 (See Appendix A for details)
4. Creatinine Clearance≥60 ml/min
5. Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN). Serum bilirubin and alkaline phosphatase ≤3x x ULN, or considered not clinically significant (e.g. Gilbert's or indirect hyperbilirubinemia) or felt to be due to underlying disease.
6. Without evidence of active acute or chronic graft versus host disease (GVHD)
7. Off all immunosuppression and corticosteroids (other than replacement dose steroids defined as equivalent to a maximum of 10 mg Prednisone daily) for ≥28 days from first treatment.
8. Off all disease targeted treatments for ≥10 days to first treatment day
9. Able to provide written informed consent
10. Women of child-bearing potential and men must agree to use adequate contraception for the duration of study participation and for 120 days after the last treatment with nivolumab.
11. No FDA approved, more appropriate therapies available for disease control as determined by the treating physician

Exclusion Criteria

1. Positive beta-human chorionic gonadotropin (HCG) in female of child-bearing potential
2. Cluster of differentiation 3 (CD3) donor chimerism <5% within 4 weeks of starting study treatment
3. Prior administration of donor lymphocyte infusion post-allogeneic transplant within the last 6 months of study treatment
4. History of or active autoimmune disease, or other syndrome that requires systemic steroids.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab.
6. Uncontrolled or active infections on treatment
7. Confirmed active human immunodeficiency virus (HIV), Hepatitis B or C infection.
8. Presence of ≥grade 3 non-hematologic toxicities as per CTCAE version 5 from any previous treatment unless it is felt to be due to underlying disease.
9. Concurrent use of investigational therapeutic agents or enrollment on another therapeutic clinical trial at any institution.

   a. Minimum of 4 weeks from last dose of investigational agent
10. Prior exposure to PD-1 or CTLA4 antibodies in the post-allogeneic transplant setting. Participants who received such agents pre-allogeneic transplant will NOT be excluded.
11. Prior exposure to daratumumab in the post-allogeneic transplant setting within two months of start date of treatment with this investigational protocol. Participants who received this agent pre-allogeneic transplant will NOT be excluded
12. Concurrent therapies targeted at disease relapse. However, previous treatments for relapsed disease are allowed.
13. Concurrent active malignancy (exceptions: treated solid malignancy in >2 years' remission, treated basal or squamous cell carcinomas of the skin)
14. History of Crohn's disease or ulcerative colitis
15. History of demyelinating disorder
16. Prior intolerance or allergy to tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated Dose | Up to 4 weeks after last dose of study treatment (approximately 3 months)
  Determine the safety and the maximum tolerated dose among two candidate doses of nivolumab in combination with tocilizumab for treatment of relapsed hematological malignancy post-allogeneic transplant. Maximum-tolerated dose is based on the determination of dose-limiting toxicities.

SECONDARY OUTCOMES:
Response Rates Based on Imaging | End of study treatment (approximately 2 months)
  The number of subjects with stable disease as evidenced by imaging (Diagnostic positron emission tomography (PET)-CT scans or CT of the neck, chest, abdomen, and pelvis).
Response Rates Based on Pathologic Response | End of study treatment (approximately 2 months)
  The number of subjects with bone marrow response (achievement of complete response; <5% blasts; stable disease; progressive disease).
Overall Survival | Up to 1 year from beginning of treatment
  The number of participants alive.
Progression-Free Survival | Up to 1 year from beginning of treatment
  Determine the number of subjects alive and in remission after treatment.
Duration of response in responding participants | Up to 1 year from the beginning of treatment
  Number of subjects with complete response or stable disease.
Dose-limiting toxicities | Up to 4 weeks after last dose of study treatment (approximately 3 months)
  The number of subjects with dose-limiting toxicities. This will be measured by the number of adverse events as defined by the NCI CTCAE version 4.03 non-hematologic ≥ grade 3-5 signs/symptoms or by the development of steroid refractory grade 2-4 graft-versus-host disease or severe chronic graft-versus-host disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No